CLINICAL TRIAL: NCT05741398
Title: Evaluation of the Efficacy and Safety of Optical System in the Treatment of - Dry Eye Disease (DED) Pilot Study
Brief Title: Evaluation of Optical System in the Treatment of - Dry Eye Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Demaod Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLN 0100
Record Dates: First submitted 2023-02-14; First posted 2023-02-23 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-02

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: Single-center, Prospective, Open Label, with Before-After Study Design
Masking Description: no masking during this study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Demaod VR system tratment (Experimental): Non-invasive light pulse generated by a non-contacting device for treating the symptoms of dry eyes and MDG.
  Interventions: Device: VR system by Demaod

INTERVENTIONS:
Device: VR system by Demaod — non-invasive light pulse generated by a non-contacting device for the treatment of the symptoms of dry eyes and MDG

SUMMARY:
Single-center, Prospective, Open Label, with Before-After Study Design, to evaluate the safety and efficacy of the optical system in the treatment of dry eye disease.

DETAILED DESCRIPTION:
Single-center, Prospective, Open Label, with Before-After Study Design. Up to 15 subjects will be enrolled in the study to provide at least 10 evaluable subjects.

All subjects will undergo 3 treatments two weeks apart (2 weeks (+/-3 days) from the previous treatment).

Follow-up visits after the last treatment visit: 4 weeks (±7 days), 12 weeks (±7 days).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older of any gender or race.
* Provide written informed consent before study participation.
* Willingness and ability to return for all study visits.
* Ocular Surface Disease Index (OSDI) questionnaire and a score of ≥ 23 at the baseline visit.
* Tear break-up time (TBUT) <10 seconds in both eyes.
* Agreement/ability to abstain from dry eye/MGD medications for the time between the treatment visit/s and the final study visit. Ocular lubricants are allowed if no changes are made during the study.

Exclusion:

* History of ocular surgery including intraocular, oculoplastic, corneal or refractive surgery within 1 year.
* Patients with giant papillary conjunctivitis.
* Patients with punctal plugs or who have had punctal cautery.
* Ocular injury or trauma, chemical burns, or limbal stem cell deficiency within 3 months of the baseline examination.
* Active ocular herpes zoster or simplex of eye or eyelid or a history of these within the last 3 months.
* Aphakic Patients.
* Cicatricial lid margin disease identified via slit lamp examination, including pemphigoid, symblepharon, etc.
* Active ocular infection (e.g., viral, bacterial, mycobacterial, protozoan, or fungal infection of the cornea, conjunctiva, lacrimal gland, lacrimal sac, or eyelids including a hordeolum or stye).
* Active ocular inflammation or history of chronic, recurrent ocular inflammation within 3 months (e.g., retinitis, macular inflammation, choroiditis, uveitis, iritis, scleritis, episcleritis, keratitis).

Criteria:

-

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
4 weeks TBUT change from baseline | up to 4 weeks post last treatment
  Change from baseline to the 4-week follow-up exam in Tear Break Up Times (TBUT), as assessed by a rater.

SECONDARY OUTCOMES:
OSDI changes from baseline to 4 and 12 weeks FU | up to 12 weeks post last treatment
  Change from baseline in patient symptoms using Ocular Surface Disease Index (OSDI) at 4-weeks and 12-weeks follow-up exam.
12 weeks TBUT change from baseline | 12 weeks post last treatment
  Changes from baseline to the 12-week follow-up exam in Tear Break Up Times (TBUT), as assessed by a rater.

CONTACTS AND LOCATIONS:
Locations (1):
- Haemek Medical Center, Afula, Israel

IPD SHARING:
Plan to Share IPD: Undecided